CLINICAL TRIAL: NCT03096288
Title: Impact of the PCSK9 Inhibitor Evolocumab on the Pharmacodynamic Effects of Clopidogrel in Patients With Atherosclerotic Cardiovascular Disease and High On-Treatment Platelet Reactivity
Brief Title: Impact of Evolocumab on the Effects of Clopidogrel in Patients With High On-Treatment Platelet Reactivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIS AMG001
Record Dates: First submitted 2017-03-23; First posted 2017-03-30 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab (Experimental): Evolocumab (Repatha) 420 mg s.c. single injection
  Interventions: Drug: Evolocumab
- Placebo (Placebo Comparator): 0.9% sodium chloride s.c. single injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Evolocumab — Patients will be randomly assigned to receive a single dose of either evolocumab 420 mg s.c. or placebo (0.9% sodium chloride s.c. injection).
  Other Names: Repatha
  Arms: Evolocumab
Other: Placebo — Patients will be randomly assigned to receive a single dose of either evolocumab 420 mg s.c. or placebo (0.9% sodium chloride s.c. injection).
  Arms: Placebo

SUMMARY:
Clopidogrel is the most widely used P2Y12 receptor inhibitor and is the only agent of this class currently recommended in patients with stable coronary artery disease (CAD) undergoing PCI, and for the treatment of stroke or PAD. Pharmacodynamic (PD) studies have shown that approximately 30-40% of patients experience high on-treatment platelet reactivity (HPR) while receiving clopidogrel treatment. Importantly HPR status has been strongly associated with an increased risk of ischemic events. Multiple approaches have been advocated to reduce HPR rates. In a previous study treatment with high-dose atorvastatin in addition to double-dose clopidogrel reduced platelet reactivity significantly more than double-dose clopidogrel alone in statin-naïve patients with stable CAD and HPR. To date, the exact biological mechanisms involved in the statin modulation of platelet function are not fully understood, although likely attributed to both its lipid-lowering and non-lipid-related effects.

Evolocumab is a monoclonal antibody targeting proprotein convertase subtilisin/kexin type 9 (PCSK9). The use of evolocumab plus standard therapy, as compared with standard therapy alone, significantly reduced the incidence of cardiovascular events. Whether the reduction in cardiovascular events is simply due to LDL reduction or might be related to other mechanisms is currently subject of investigation. Although LDL reduction with statin therapies has been associated with reduction in platelet reactivity, to date the effects on platelet aggregation of adjunctive lipid lowering with evolocumab has not been explored.

The aim of the present study is to investigate the effects of evolocumab in addition to statin therapy on HPR rates and platelet reactivity in patients with atherosclerotic cardiovascular disease (ASCVD) and HPR while on clopidogrel treatment.

DETAILED DESCRIPTION:
Clopidogrel is the most widely used P2Y12 receptor inhibitor and is the only agent of this class currently recommended in patients with stable coronary artery disease (CAD) undergoing PCI, and for the treatment of stroke or PAD. Although the efficacy of DAPT with aspirin and clopidogrel has been consistently shown in different clinical settings, rates of ischemic recurrences remain elevated despite this treatment regimen, especially in high risk patients. This has been in part attributed to the high interindividual variability in responses to clopidogrel. Pharmacodynamic (PD) studies have shown that approximately 30-40% of patients experience high on-treatment platelet reactivity (HPR) while receiving clopidogrel treatment. Importantly HPR status has been strongly associated with an increased risk of ischemic events, in particular stent thrombosis, in patients with ACS and following PCI. This underscores the need for strategies aimed to reduce HPR rates in patients treated with clopidogrel. Multiple approaches have been advocated to reduce HPR rates. The pleiotropic effects associated with lipid lowering therapies, in particular statins, have been subject to extensive research. In a previous study treatment with high-dose atorvastatin in addition to double-dose clopidogrel reduced platelet reactivity significantly more than double-dose clopidogrel alone in statin-naïve patients with stable CAD and HPR. To date, the exact biological mechanisms involved in the statin modulation of platelet function are not fully understood, although likely attributed to both its lipid-lowering and non-lipid-related effects.

Evolocumab is a monoclonal antibody targeting proprotein convertase subtilisin/kexin type 9 (PCSK9) that is administered subcutaneously (s.c.) at a dosage of 140 mg every 2 weeks or 420 mg once monthly. In clinical trials evolocumab was more effective than placebo and/or ezetimibe in reducing LDL cholesterol, including when added to statin therapy. The use of evolocumab plus standard therapy, as compared with standard therapy alone, significantly reduced the incidence of cardiovascular events. Whether the reduction in cardiovascular events is simply due to LDL reduction or might be related to other mechanisms is currently subject of investigation. Although LDL reduction with statin therapies has been associated with reduction in platelet reactivity, to date the effects on platelet aggregation of adjunctive lipid lowering with evolocumab has not been explored.

The aim of the present study is to investigate the effects of evolocumab in addition to statin therapy on HPR rates and platelet reactivity in patients with atherosclerotic cardiovascular disease (ASCVD) and HPR while on clopidogrel treatment.

ELIGIBILITY:
Inclusion criteria:

1. Patients with atherosclerotic cardiovascular disease (ASCVD), defined as prior ACS, history of myocardial infarction, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack, or PAD presumed to be of atherosclerotic origin.
2. On therapy with clopidogrel (75mg od), with or without low-dose aspirin (81mg od), as per standard-of-care for at least 30 days.
3. HPR, defined as P2Y12 reaction units (PRU) > 208 by VerifyNow P2Y12.
4. Fasting LDL-cholesterol ≥70 mg/dL or a non-high-density lipoprotein cholesterol (HDL-C) of ≥100 mg/dL after ≥2 weeks of optimized stable lipid-lowering therapy with maximally tolerated dose of statin, which would ideally include a high-intensity statin, but must be at least moderate intensity statin (i.e. atorvastatin 20 mg or equivalent, with or without ezetimibe. Maximal tolerated dose will be defined based on patient clinical history (no statin re-challenge will be performed).
5. Age ≥ 18 years old.

Exclusion criteria:

1. On treatment with any oral anticoagulant (vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxaban).
2. On treatment with any antiplatelet agent other than aspirin and clopidogrel in the past 14 days.
3. Use of PCSK9 inhibitors in the past 90 days
4. Creatinine clearance <30 mL/minute.
5. Known severe hepatic impairment.
6. History of a serious hypersensitivity reaction to evolocumab
7. Hemodynamic instability
8. Pregnant and breastfeeding women [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Ortega-Paz L, Rollini F, Been L, Rivas A, Maaliki N, Zhou X, Pineda AM, Suryadevara S, Soffer D, Zenni M, Angiolillo DJ. Impact of evolocumab on the pharmacodynamic profiles of clopidogrel in patients with atherosclerotic cardiovascular disease: a randomised, double-blind, placebo-controlled study. EuroIntervention. 2023 Mar 20;18(15):1254-1265. doi: 10.4244/EIJ-D-22-00719. PMID 36602868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between October 2017 and May 2020 at the University of Florida Health Science Center at UF Health Jacksonville - Division of Cardiology
Pre-assignment Details: 259 patients were consented to participate in the study. Of these, 165 were screen failures and 10 withdrew consent before randomization. Thus, 84 patients were randomized and received study treatment.
Groups:
- HPR - Evolocumab; HPR - Placebo: Patients with high platelet reactivity (HPR) will be randomly assigned to receive a single dose of either evolocumab 420 mg s.c. or placebo (0.9% sodium chloride s.c. injection).
- NPR - Evolocumab; NPR - Placebo: Patients with normal platelet reactivity (NPR) will be randomly assigned to receive a single dose of either evolocumab 420 mg s.c. or placebo (0.9% sodium chloride s.c. injection).
Period: Overall Study
Arm/Group | HPR - Evolocumab | HPR - Placebo | NPR - Evolocumab | NPR - Placebo
Started | 19 | 18 | 22 | 25
Completed | 19 | 17 | 22 | 24
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HPR - Evolocumab | HPR - Placebo | NPR - Evolocumab | NPR - Placebo | Total
Number analyzed (Participants) | 19 | 18 | 22 | 25 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8) | 62 (8) | 63 (8) | 58 (8) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 10 | 8 | 32
  Male | 11 | 12 | 12 | 17 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 10 | 11 | 10 | 46
  White | 4 | 7 | 11 | 14 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 107 (29) | 109 (42) | 91 (30) | 99 (31) | 101 (33)

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Defined by VerifyNow PRU in HPR and NPR Patients
Description: The primary end point of our study is the comparison of P2Y12 reaction units (PRU) measured by VerifyNow between evolocumab and placebo at 30 days after randomization. PRU is a well-established measure of platelet reactivity and aggregation in response to antiplatelet medications. The higher is the PRU the lower is the effect of the antiplatelet medication. HPR is defined as PRU>208 and NPR as PRU 85-208.
Time Frame: 30 days
Population: Patient with valid data at 30 days were analyzed
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | HPR - Evolocumab | HPR - Placebo | NPR - Evolocumab | NPR - Placebo
Number analyzed (Participants) | 19 | 17 | 22 | 24
PRU | 219 (38) | 241 (52) | 141 (54) | 159 (41)
Statistical Analysis 1: Comparison: HPR - Evolocumab vs HPR - Placebo; Test type: Superiority; p = 0.169, t-test, 2 sided; Mean Difference (Final Values) = 22, 95% CI 2-sided [-9 to 52]
Statistical Analysis 2: Comparison: NPR - Evolocumab vs NPR - Placebo; Test type: Superiority; p = 0.236, t-test, 2 sided; Median Difference (Final Values) = 17, 95% CI 2-sided [-11 to 45]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Non serious adverse events are reported only if frequency >5%.
Groups:
- HPR - Evolocumab; NPR - Evolocumab: Evolocumab (Repatha) 420 mg s.c. single injection
  Evolocumab: Patients will be randomly assigned to receive a single dose of either evolocumab 420 mg s.c. or placebo (0.9% sodium chloride s.c. injection).
- HPR - Placebo; NPR - Placebo: 0.9% sodium chloride s.c. single injection
  Placebo: Patients will be randomly assigned to receive a single dose of either evolocumab 420 mg s.c. or placebo (0.9% sodium chloride s.c. injection).
Arm/Group | HPR - Evolocumab | HPR - Placebo | NPR - Evolocumab | NPR - Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/22 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/18 | 1/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/22 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPR - Evolocumab (N=19) | HPR - Placebo (N=18) | NPR - Evolocumab (N=22) | NPR - Placebo (N=25)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03096288/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03096288/ICF_001.pdf